CLINICAL TRIAL: NCT04770649
Title: VOICES: Vaccine Observation to Include All Communities for Equitable Science
Brief Title: Vaccine Observation to Include All Communities for Equitable Science
Acronym: VOICES
Status: Terminated | Type: Observational
Why Stopped: No longer of interest to the company
Sponsor: Persephone Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: PB-2021-01
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2021-02

CONDITIONS: Vaccine Response Impaired; Vaccine Adverse Reaction
Keywords: SARS-CoV-2; COVID-19; gut microbiome; vaccine
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COVID-19 vaccine recipients: Subjects who have an appointment to receive a COVID-19 vaccine, and are able to provide samples prior to and after their first vaccine dose.
  Interventions: Biological: COVID-19 vaccine

INTERVENTIONS:
Biological: COVID-19 vaccine — Any vaccine for COVID-19

SUMMARY:
VOICES is a longitudinal, prospective, observational study that will enroll up to 10,000 subjects of diverse racial backgrounds being administered an emergency use authorized COVID-19 vaccine, for collection and analysis of stool and blood samples. It has recently been shown that the gut microbiome, the collection of microbes that line our GI tract, play a significant role in vaccine immune response and severe complications from COVID-19. The identification of biomarkers may aid in predicting response to vaccination and are critical towards improving vaccine-induced immunity. These real-world patient derived biomarkers could be used as interventional targets for the design of innovative adjuvant co-therapies that can boost an effective immune response to the vaccine, enhancing efficacy for a broader population, including those at most risk.

Subjects who meet the entry criteria will provide two samples each of blood, one prior to and one following vaccine administration. Follow-up questionnaires will be sent at 3, 6, 9, and 12 months to determine if participants have contracted COVID-19 or have experienced any adverse effects of the vaccine. Nasal swab samples will also be collected from participants that have contracted COVID-19. The samples will be analyzed to determine the impact of gut microbiome composition and function on the immune system and vaccine efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Men or women who are ≥ 18 years old and expecting to receive the SARS-CoV-2 vaccine within the next 30 days.
* Subjects who are able to provide written informed consent.

Exclusion Criteria:

* Subjects with known HIV, Hepatitis A, Hepatitis B, Hepatitis C, or SARS-CoV-2 infection within 4 weeks of vaccination
* Subjects without the mental capacity to complete either a written or online questionnaire, alone or with assistance, or make sound decisions
* Women who are pregnant, plan on becoming pregnant, or are nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It is anticipated that 10,000 subjects will be enrolled in this study. It is preferred that enrollment is balanced by sex; however, it is not required. All efforts will be made to provide racial/ethnic balance, with a goal of 50% underrepresented minorities.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Determine whether the microbiome composition can predict effectiveness of vaccine. | 6-12 months
  Whole genome sequencing and metabolomics will be used to characterize the patient's microbiome, and whether there is any correlation with subjects who contract COVID-19 post-vaccination

SECONDARY OUTCOMES:
Identify correlations between microbiome composition and immune system response to the vaccine | 3-6 months
  Immune cell profile and cytokine analysis will be performed on the blood samples to characterize the patient's immune phenotype, and determine how it correlates to microbiome composition
Track coronavirus variants of any individuals infected | 6-12 months
  Any subject who contracts COVID-19 after vaccination will provide a nasal swab, which will be subject to viral sequencing to determine whether vaccinated individuals are more susceptible to certain variants
Build a library of samples and data for future research | 6-24 months
  Samples will be stored and data saved in a HIPAA-compliant database. Samples will be linked to patient metadata

CONTACTS AND LOCATIONS:
Locations (1):
- Persephone Biosciences, Inc., San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No